CLINICAL TRIAL: NCT03038997
Title: Early Detection of Cardiac Toxicity in Childhood Cancer Survivors
Status: Terminated | Type: Observational
Why Stopped: IRB approval expired
Sponsor: Niti Dham (Other)
Responsible Party: Sponsor-Investigator, Niti Dham, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 5405
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure; Cardiotoxicity
MeSH Terms: conditions — Heart Failure; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood specimen equal to 1 teaspoonful will be collected for future analysis to be used to identify serum biomarkers in myocardial fibrosis, and to validate the potential use for diagnostic purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate cardiac MRI and/or serum biomarkers for detecting cardiac cardiac toxicity in children who received anthracycline based chemotherapy (ABC).

DETAILED DESCRIPTION:
Cardiac toxicity is a significant potential complication for patients receiving anthracycline chemotherapy. Cells in the cardiovascular system have limited regenerative capability, making them susceptible to long term adverse effects from these chemotherapeutic agents. The ability to detect subclinical changes in cardiac function will allow clinicians to use proven treatments to prevent further progression in this vulnerable population. The current standard testing uses echocardiography, which is not as sensitive as cardiac MRI or serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have received anthracycline based chemotherapy
* Age: 8 years old - 25 years old
* Subjects that do not require sedation for cardiac MRI.
* Subjects must have completed treatment in the last 10 years

Exclusion Criteria:

* Patients with significant congenital heart defects
* Patients with renal injury or renal failure, defined as an estimated glomerular filtration rate [eGFR] <30 ml/min/1.73 m2 body surface area), as previously calculated)
* Patients that require sedation for a cardiac MRI
* Subjects that are pregnant or lactating
* Patients with contraindications to a cardiac MRI:
* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Neural stimulator
* Metallic ocular foreign body
* Any implanted device (i.e. insulin pump, drug infusion device)
* Claustrophobia
* Metal shrapnel or bullet
* Investigator assessment of inability to comply with protocol
* Unable/unwilling to lie still throughout the research procedure
* Persons with cognitive impairment

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with previous exposure to anthracyclines between the ages of 8-25 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Echocardiogram marker measurements pre ABC chemo and post ABC | At the end of each cardiac MRI exam through study completion, up to 5 years
  •Measure echocardiogram markers on pre anthracycline based chemotherapy (ABC) and post ABC echocardiograms, using standard echocardiogram measurements and speckle tracking.

SECONDARY OUTCOMES:
Detection of cardiac toxicity on MRI and echocardiogram | At the end of each cardiac MRI exam through study completion, up to 5 years
  •Measure sensitivity of detecting cardiac toxicity between standard echocardiogram, speckle tracking on echo, and MRI
Serum biomarkers correlation | At the end of the study, up to 10 years
  •Correlate measurement of serum biomarkers with prevalence of cardiac changes measured on echocardiograms and MRI imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Niti Dham, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz RG, Jain D, Storozynsky E. Traditional and novel methods to assess and prevent chemotherapy-related cardiac dysfunction noninvasively. J Nucl Cardiol. 2013 Jun;20(3):443-64. doi: 10.1007/s12350-013-9707-1. PMID 23572315
- [Background] Lipshultz SE, Adams MJ, Colan SD, Constine LS, Herman EH, Hsu DT, Hudson MM, Kremer LC, Landy DC, Miller TL, Oeffinger KC, Rosenthal DN, Sable CA, Sallan SE, Singh GK, Steinberger J, Cochran TR, Wilkinson JD; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Basic Cardiovascular Sciences, Council on Cardiovascular and Stroke Nursing, Council on Cardiovascular Radiolo. Long-term cardiovascular toxicity in children, adolescents, and young adults who receive cancer therapy: pathophysiology, course, monitoring, management, prevention, and research directions: a scientific statement from the American Heart Association. Circulation. 2013 Oct 22;128(17):1927-95. doi: 10.1161/CIR.0b013e3182a88099. Epub 2013 Sep 30. No abstract available. PMID 24081971
- [Background] Kremer LC, van Dalen EC, Offringa M, Voute PA. Frequency and risk factors of anthracycline-induced clinical heart failure in children: a systematic review. Ann Oncol. 2002 Apr;13(4):503-12. doi: 10.1093/annonc/mdf118. PMID 12056699
- [Background] Kremer LC, van der Pal HJ, Offringa M, van Dalen EC, Voute PA. Frequency and risk factors of subclinical cardiotoxicity after anthracycline therapy in children: a systematic review. Ann Oncol. 2002 Jun;13(6):819-29. doi: 10.1093/annonc/mdf167. PMID 12123328
- [Background] Shankar SM, Marina N, Hudson MM, Hodgson DC, Adams MJ, Landier W, Bhatia S, Meeske K, Chen MH, Kinahan KE, Steinberger J, Rosenthal D; Cardiovascular Disease Task Force of the Children's Oncology Group. Monitoring for cardiovascular disease in survivors of childhood cancer: report from the Cardiovascular Disease Task Force of the Children's Oncology Group. Pediatrics. 2008 Feb;121(2):e387-96. doi: 10.1542/peds.2007-0575. Epub 2008 Jan 10. PMID 18187811
- [Background] Steinherz LJ, Graham T, Hurwitz R, Sondheimer HM, Schwartz RG, Shaffer EM, Sandor G, Benson L, Williams R. Guidelines for cardiac monitoring of children during and after anthracycline therapy: report of the Cardiology Committee of the Childrens Cancer Study Group. Pediatrics. 1992 May;89(5 Pt 1):942-9. PMID 1579408
- [Background] Cheung YF, Hong WJ, Chan GC, Wong SJ, Ha SY. Left ventricular myocardial deformation and mechanical dyssynchrony in children with normal ventricular shortening fraction after anthracycline therapy. Heart. 2010 Jul;96(14):1137-41. doi: 10.1136/hrt.2010.194118. Epub 2010 May 29. PMID 20511624
- [Background] Mavinkurve-Groothuis AM, Marcus KA, Pourier M, Loonen J, Feuth T, Hoogerbrugge PM, de Korte CL, Kapusta L. Myocardial 2D strain echocardiography and cardiac biomarkers in children during and shortly after anthracycline therapy for acute lymphoblastic leukaemia (ALL): a prospective study. Eur Heart J Cardiovasc Imaging. 2013 Jun;14(6):562-9. doi: 10.1093/ehjci/jes217. Epub 2012 Oct 29. PMID 23109647
- [Background] Lunning MA, Kutty S, Rome ET, Li L, Padiyath A, Loberiza F, Bociek RG, Bierman PJ, Vose JM, Armitage JO, Porter TR. Cardiac magnetic resonance imaging for the assessment of the myocardium after doxorubicin-based chemotherapy. Am J Clin Oncol. 2015 Aug;38(4):377-81. doi: 10.1097/COC.0b013e31829e19be. PMID 24192805
- [Background] Weidemann F, Jamal F, Sutherland GR, Claus P, Kowalski M, Hatle L, De Scheerder I, Bijnens B, Rademakers FE. Myocardial function defined by strain rate and strain during alterations in inotropic states and heart rate. Am J Physiol Heart Circ Physiol. 2002 Aug;283(2):H792-9. doi: 10.1152/ajpheart.00025.2002. PMID 12124229
- [Background] Pirat B, McCulloch ML, Zoghbi WA. Evaluation of global and regional right ventricular systolic function in patients with pulmonary hypertension using a novel speckle tracking method. Am J Cardiol. 2006 Sep 1;98(5):699-704. doi: 10.1016/j.amjcard.2006.03.056. Epub 2006 Jul 17. PMID 16923465
- [Background] Dogru A, Cabuk D, Sahin T, Dolasik I, Temiz S, Uygun K. Evaluation of cardiotoxicity via speckle-tracking echocardiography in patients treated with anthracyclines. Onkologie. 2013;36(12):712-6. doi: 10.1159/000356850. Epub 2013 Nov 20. PMID 24356562
- [Background] Sawaya H, Sebag IA, Plana JC, Januzzi JL, Ky B, Tan TC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Assessment of echocardiography and biomarkers for the extended prediction of cardiotoxicity in patients treated with anthracyclines, taxanes, and trastuzumab. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):596-603. doi: 10.1161/CIRCIMAGING.112.973321. Epub 2012 Jun 28. PMID 22744937
- [Background] Wassmuth R, Lentzsch S, Erdbruegger U, Schulz-Menger J, Doerken B, Dietz R, Friedrich MG. Subclinical cardiotoxic effects of anthracyclines as assessed by magnetic resonance imaging-a pilot study. Am Heart J. 2001 Jun;141(6):1007-13. doi: 10.1067/mhj.2001.115436. PMID 11376317
- [Background] Oberholzer K, Kunz RP, Dittrich M, Thelen M. [Anthracycline-induced cardiotoxicity: cardiac MRI after treatment for childhood cancer]. Rofo. 2004 Sep;176(9):1245-50. doi: 10.1055/s-2004-813416. German. PMID 15346258
- [Background] Kellman P, Wilson JR, Xue H, Bandettini WP, Shanbhag SM, Druey KM, Ugander M, Arai AE. Extracellular volume fraction mapping in the myocardium, part 2: initial clinical experience. J Cardiovasc Magn Reson. 2012 Sep 11;14(1):64. doi: 10.1186/1532-429X-14-64. PMID 22967246
- [Background] Florian A, Ludwig A, Rosch S, Yildiz H, Sechtem U, Yilmaz A. Myocardial fibrosis imaging based on T1-mapping and extracellular volume fraction (ECV) measurement in muscular dystrophy patients: diagnostic value compared with conventional late gadolinium enhancement (LGE) imaging. Eur Heart J Cardiovasc Imaging. 2014 Sep;15(9):1004-12. doi: 10.1093/ehjci/jeu050. Epub 2014 Mar 30. PMID 24686257
- [Background] Mahrholdt H, Wagner A, Judd RM, Sechtem U, Kim RJ. Delayed enhancement cardiovascular magnetic resonance assessment of non-ischaemic cardiomyopathies. Eur Heart J. 2005 Aug;26(15):1461-74. doi: 10.1093/eurheartj/ehi258. Epub 2005 Apr 14. PMID 15831557
- [Background] Menon SC, Etheridge SP, Liesemer KN, Williams RV, Bardsley T, Heywood MC, Puchalski MD. Predictive value of myocardial delayed enhancement in Duchenne muscular dystrophy. Pediatr Cardiol. 2014 Oct;35(7):1279-85. doi: 10.1007/s00246-014-0929-z. Epub 2014 May 15. PMID 24830760
- [Background] Yildirim A, Tunaoglu FS, Kambur K, Pinarli FG. The utility of NT-proBNP and various echocardiographic methods in the determination of doxorubicin induced subclinical late cardiotoxicity. Kardiol Pol. 2013;71(1):40-6. PMID 23348532
- [Background] Colombo A, Cardinale D. Using cardiac biomarkers and treating cardiotoxicity in cancer. Future Cardiol. 2013 Jan;9(1):105-18. doi: 10.2217/fca.12.73. PMID 23259478
- [Background] Ky B, Putt M, Sawaya H, French B, Januzzi JL Jr, Sebag IA, Plana JC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Early increases in multiple biomarkers predict subsequent cardiotoxicity in patients with breast cancer treated with doxorubicin, taxanes, and trastuzumab. J Am Coll Cardiol. 2014 Mar 4;63(8):809-16. doi: 10.1016/j.jacc.2013.10.061. Epub 2013 Nov 27. PMID 24291281
- [Background] Lai WW, Geva T, Shirali GS, Frommelt PC, Humes RA, Brook MM, Pignatelli RH, Rychik J; Task Force of the Pediatric Council of the American Society of Echocardiography; Pediatric Council of the American Society of Echocardiography. Guidelines and standards for performance of a pediatric echocardiogram: a report from the Task Force of the Pediatric Council of the American Society of Echocardiography. J Am Soc Echocardiogr. 2006 Dec;19(12):1413-30. doi: 10.1016/j.echo.2006.09.001. No abstract available. PMID 17138024
- [Background] Ugander M, Oki AJ, Hsu LY, Kellman P, Greiser A, Aletras AH, Sibley CT, Chen MY, Bandettini WP, Arai AE. Extracellular volume imaging by magnetic resonance imaging provides insights into overt and sub-clinical myocardial pathology. Eur Heart J. 2012 May;33(10):1268-78. doi: 10.1093/eurheartj/ehr481. Epub 2012 Jan 24. PMID 22279111
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423
- [Background] Cao Y, Huang DQ, Shih G, Prince MR. Signal Change in the Dentate Nucleus on T1-Weighted MR Images After Multiple Administrations of Gadopentetate Dimeglumine Versus Gadobutrol. AJR Am J Roentgenol. 2016 Feb;206(2):414-9. doi: 10.2214/AJR.15.15327. Epub 2015 Dec 23. PMID 26700156
- [Background] Jost G, Lenhard DC, Sieber MA, Lohrke J, Frenzel T, Pietsch H. Signal Increase on Unenhanced T1-Weighted Images in the Rat Brain After Repeated, Extended Doses of Gadolinium-Based Contrast Agents: Comparison of Linear and Macrocyclic Agents. Invest Radiol. 2016 Feb;51(2):83-9. doi: 10.1097/RLI.0000000000000242. PMID 26606548